CLINICAL TRIAL: NCT01142063
Title: A Single Dose Bioequivalence Study Comparing The Commercial Tablet Formulation To The Clinical Tablet Of Neratinib In Healthy Subjects
Brief Title: A Single Dose Bioequivalence Study Of Neratinib In Healthy Subjects
Status: Completed | Type: Observational
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: B1891021; 3144A1-1127
Record Dates: First submitted 2010-06-09; First posted 2010-06-11 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: Neratinib
MeSH Terms: interventions — neratinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Treatment A (Reference fasted): Treatment A (Reference fasted): A 40 mg tablet strength neratinib administered as a single dose of 6 x 40 mg under fasted condition.
  Interventions: Drug: Neratinib
- Treatment B (Test fasted): Treatment B (Test fasted): A 240 mg tablet strength neratinib administered as a single dose of 1 x 240 mg under fasted condition.
  Interventions: Drug: Neratinib
- Treatment C (Reference fed): Treatment C (Reference fed): A 40 mg tablet strength neratinib administered as a single dose of 6 x 40 mg under fed condition.
  Interventions: Drug: Neratinib
- Treatment D (Test fed): Treatment D (Test fed): A 240 mg tablet strength neratinib administered as a single dose of 1 x 240 mg under fed condition.
  Interventions: Drug: Neratinib

INTERVENTIONS:
Drug: Neratinib — Tablet, a 240 mg single oral dose
  Other Names: HKI-272
  Groups: Treatment A (Reference fasted)
Drug: Neratinib — Tablet, a 240 mg single oral dose
  Other Names: HKI-272
  Groups: Treatment B (Test fasted)
Drug: Neratinib — Tablet, a 240 mg single oral dose
  Other Names: HKI-272
  Groups: Treatment C (Reference fed)
Drug: Neratinib — Tablet, a 240 mg single oral dose
  Other Names: HKI-272
  Groups: Treatment D (Test fed)

SUMMARY:
The purpose of the study is to demonstrate the bioequivalence of the proposed commercial neratinib tablet formulation (240 mg strength x 1) to the reference Phase 3 tablet formulation (40 mg tablet strength x 6) under fed and fasted conditions in healthy subjects.

DETAILED DESCRIPTION:
The study will be an open label, randomized, 4 period, 4 treatment, 4 sequence (Williams design), cross over.

ELIGIBILITY:
Inclusion Criteria:

* An informed consent document signed and dated by the subject or a legally acceptable representative.
* Healthy male and/or female of non-childbearing potential subjects between the ages of 18 and 55 years, inclusive (healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG, and clinical laboratory tests).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Cohorts will be selected from healthy volunteers.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) and Area under the plasma concentration-time profile from time zero extrapolated to infinite time for neratinib (AUCinf) | 0 to 48 hour post-dose

SECONDARY OUTCOMES:
Plasma Time for Cmax (Tmax), Area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration (Clast) (AUClast) and Terminal elimination half-life (t1/2) for neratinib | 0 to 48 hour post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Puma, Study Director — Biotechnology
Locations (1):
- Investigational Site, New Haven, Connecticut, United States